CLINICAL TRIAL: NCT07207590
Title: The Effect of Gamification-Based Instructional Design Developed for Postpartum Hemorrhage Management on Knowledge Acquisition and Retention
Brief Title: The Effect of Gamification-Based Instructional Design Developed
Acronym: PPH-GamEd
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Zeynep Seyyide KAYA, Research Assistant, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 148-KARAR 31-4.10.2024; 148-KARAR 31-4.10.2024 (Other: Cukuruva University)
Record Dates: First submitted 2025-09-19; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Midwifery Student
Keywords: Postpartum hemorrhage; Midwife; Learning; Motivation; Education; Student; Gamification; Game; Web application
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single-blind and stratified randomization will be performed to prevent selection bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- invervention group: midwifery student (Experimental): Gamified PPH Training
  Interventions: Other: web-based gamification application
- control group: midwifery student (Active Comparator): traditional classroom learning techniques
  Interventions: Other: control group: traditional classroom learning techniques

INTERVENTIONS:
Other: web-based gamification application — Subject review and case analysis will be performed through a web-based gamification application on postpartum hemorrhage management, which will be prepared and developed by the game developer.
  Other Names: intervention group
  Arms: invervention group: midwifery student
Other: control group: traditional classroom learning techniques — Students in the control group will be taught topic review and case analysis using traditional classroom learning techniques
  Arms: control group: midwifery student

SUMMARY:
Turkish)

Abstract:

Purpose: Considering the importance of postpartum hemorrhage management in reducing preventable maternal deaths and the key role midwives play in providing this care, it is important to increase the knowledge and skills of midwifery students in this area. Many educational curricula offer weekly or semester-long courses. The Ministry also provides post-graduation training. However, considering the rates and causes of maternal deaths, it is thought that there are limitations regarding the retention of this topic. Studies on gamification in different fields and topics demonstrate its positive impact on knowledge retention. The research aims to examine the impact of a technology-based educational intervention using gamification to support midwifery students' learning and retention of knowledge on postpartum hemorrhage management.

Materials and Methods: The research will be conducted as a randomized controlled experimental study. The research population will consist of all students enrolled in the Midwifery Program in the 2024-2026 academic year, and the sample will consist of 4th-year Midwifery undergraduate students. The study sample will consist of all students in their fourth year and have completed their course registration during the 2024-2026 academic year, following the finalization of the educational content.

Single-blind, stratified randomization will be employed to prevent selection bias. A pretest, posttest, and post-study retention test will be administered during the intervention phase of the study. After data collection, the control group will receive topic review and case analysis through gamification.

After a detailed literature review for the study, educational materials will be planned per the Ministry of Health's Postpartum Care and Emergency Obstetric Care guidelines, with identical topic content for the experimental and control groups. The experimental and control groups will receive a PowerPoint presentation on postpartum hemorrhage management, prepared by the researcher, during the first week. One week later, the experimental group will receive topic review and case analysis using a web-based gamification application on postpartum hemorrhage management, developed by the researcher and the game developer. Students in the control group will receive topic review and case analysis using traditional classroom learning techniques. Expert opinions will be sought to evaluate the content created for the experimental and control groups. The pilot group will implement the content created based on expert opinions. After the pilot application, the game and educational content will be finalized based on expert opinions.

A pretest will be administered before the training, a posttest after the training and gamification application, and a retention test 3 months after the intervention. The pretest will be administered before the gamification experience and the training, the posttest after the gamification experience and the traditional method, and a retention test 3 months after the training. Data will be collected using an introductory information form and the Postpartum Hemorrhage Knowledge Test.

Data obtained from the study will be analyzed in a computer environment using TAP 6 and SPSS (Statistical Package for Social Sciences/25.0 for Windows). The study's independent variable is the gamification teaching activity developed for postpartum hemorrhage management. The dependent variable is the students' descriptive characteristics and their knowledge level about postpartum hemorrhage management. Data will be analyzed using appropriate analysis methods after performing normality tests. Contribution to Science: Using innovative learning styles to improve the quality of education has recently become popular. As new generations grow up in the constantly evolving age of technology, old, classical methods are considered inadequate. Therefore, the plan is to use a web application developed using gamification. This new trend is innovative and technology-infused, entertaining and teaching, and avoids boring and monotonous narratives. This web application aims to help midwifery students learn postpartum hemorrhage management more memorably, enhancing their knowledge and problem-solving skills. While studies on this topic are only beginning to increase in the health field, they are limited in midwifery. Considering the importance of midwives, who play a key role in postpartum hemorrhage management and provide this care in reducing preventable maternal deaths, it is crucial to increase midwifery students' knowledge and skills in this area. A new, affordable, accessible method will be developed to achieve this most effectively. This method will provide equal educational opportunities to students who teach in different cities with varying equipment levels.

DETAILED DESCRIPTION:
Materials and Methods Type and Purpose of the Study The study was planned as a randomized controlled experimental study. The purpose of the study was to evaluate the effectiveness of a technology-based educational intervention using gamification to support midwifery students' learning and retention of knowledge on postpartum hemorrhage management.

Place and Time of the Study The study will be conducted at the Midwifery Department of the Faculty of Health Sciences at Çukurova University during the 2024-2026 academic year. The planned training will be conducted outside of the curriculum, during free time available in the students' schedules, and on a weekday.

Research Population and Sample The research population will consist of all students enrolled in the Midwifery Program in the 2024-2026 academic year, and the sample will consist of fourth-year undergraduate students who completed their course registrations following the completion of the study infrastructure. The research sample will consist of all fourth-year students who completed their course registrations during the 2024-2026 academic year following the finalization of the educational content. Students from the entire sample who meet the inclusion criteria and volunteer to participate in the study will be included in the study.

Inclusion criteria:

* Volunteering to participate in the study,
* Being a 4th-year midwifery student,
* Knowing how to use a scanner,
* Having successfully completed all courses on normal and high-risk pregnancies, and normal and high-risk births.

Exclusion criteria:

- Having received any prior training on postpartum hemorrhage management, Randomization Single-blind, stratified randomization will be conducted to prevent selection bias. To ensure similar achievement levels for students in the experimental and control groups, groups will be stratified by grouping achievement levels based on the final grade lists of the courses covered in the inclusion criteria. Randomization will then be conducted via Random.org. A pretest, posttest, and post-intervention retention test will be administered during the intervention phase of the study. The pretest will be administered before the training, the posttest after the training and gamification program, and the retention test 3 months after the intervention. After data collection, the control group students will be administered a gamification-based case study. Research Implementation Procedure The primary objective of the study is to increase midwifery students' knowledge of postpartum hemorrhage management, problem-solving skills in case management, and retention of knowledge. The study will be conducted in the form of a pretest, posttest, and retention assessment test. The pretest will be administered before the training, the posttest after the training and intervention, and the retention test three months after the training and intervention. Prior to the implementation, permissions for the use of the Postpartum Care and Emergency Obstetric Care guidelines will be obtained from the Public Health Directorate and the institutional permit will be obtained from Çukurova University. A Clinical Trial Number will be obtained.

Intervention Group:

Students in the intervention group will be introduced to postpartum hemorrhage management through a PowerPoint presentation in the first week, followed by a role-playing method for reviewing the topic and performing a case study. The effectiveness of the training will be evaluated through a pretest, posttest, and retention test three months later.

Control Group: Students in the control group will be taught postpartum bleeding management using a PowerPoint presentation during the first week. The following week, they will be given a review of the topic and a case study using traditional in-class learning techniques. The effectiveness of the training will be evaluated with a pretest, posttest, and a retention test after three months.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the study
* Must be a 4th-year midwifery student
* Must know how to use a scanner
* Must have successfully completed all courses on normal and risky pregnancies and normal and risky births

Exclusion Criteria:

* Having received any prior training on postpartum hemorrhage management

Ages: 17 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — female
Enrollment: 150 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Introductory Information Form | 3 months
  This form was composed of 9 questions covering socio-demographic information prepared by the researchers in line with the literature.
Postpartum Hemorrhage Management Knowledge Test | 3 months
  This will be developed by the researcher based on the educational content developed in accordance with the postpartum hemorrhage algorithm in the Postpartum Care Guide (2018) and Emergency Obstetric Care Guide (2022), prepared by the General Directorate of Public Health of the Ministry of Health. The questions are planned to be multiple-choice problems to measure the knowledge in the training.

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 41. Ordu Y, Çalışkan N. (2021). Hemşirelik eğitiminde oyun temelli öğrenmede yenilikçi bir yaklaşım: Sanal oyun simülasyonu. JHS. 18(4):657- 664.
- [Background] Roman P, Rodriguez-Arrastia M, Molina-Torres G, Marquez-Hernandez VV, Gutierrez-Puertas L, Ropero-Padilla C. The escape room as evaluation method: A qualitative study of nursing students' experiences. Med Teach. 2020 Apr;42(4):403-410. doi: 10.1080/0142159X.2019.1687865. Epub 2019 Nov 18. PMID 31738615